# Statistical Analysis Plan (SAP)

PRISM-EXT: An Open-Label Extension of CP101 Trial Evaluating Oral Full-Spectrum Microbiota® (CP101) in Subjects with Recurrence of *Clostridium difficile* Infection

Protocol Number: CP101-CDI-E02

Investigational Product: Full-Spectrum Microbiota® (CP101)

Phase: 2 (Open-Label Study)

Protocol Version: Version 4.0, 20 December 2019

SAP Version: Version 1.0, 5 April 2021

Finch Research and Development LLC 200 Inner Belt Road, Suite 400 Somerville, MA 02143

#### **Confidentiality Statement:**

This document contains confidential information of Finch Research and Development LLC (the Sponsor) which must not be reproduced, published, or otherwise disclosed to anyone other than the recipient(s), members of the ethics committee(s) or regulatory authorities. The document and the information contained herein cannot be used for any purpose other than the evaluation or conduct of the clinical investigation described in this document without prior written approval from Finch Research and Development LLC. The foregoing shall not apply to disclosure required by applicable laws or governmental regulations. Notice must be provided to Finch Research and Development LLC of any such disclosure as soon as practicable.

#### SAP APPROVAL FORM

Document Title:

Statistical Analysis Plan

Protocol Number:

CP101-CDI-E02

Study Title:

PRISM-EXT: An Open-Label Extension of CP101 Trial Evaluating Oral

Full-Spectrum Microbiota® (CP101) in Subjects with Recurrence of

Clostridium difficile Infection

This Statistical Analysis Plan is prepared, reviewed and approved by:



# TABLE OF CONTENTS

| SAP A | PPROVAL FORM | 2 |
|--------|--------------------------------------------------|----|
| TABLI | E OF CONTENTS | 3 |
| LIST C | OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 5 |
| 1. | INTRODUCTION | 6 |
| 2. | STUDY OBJECTIVES | 6 |
| 3. | STUDY DESIGN | 6 |
| 3.1. | General Study Design and Plan | 6 |
| 3.2. | Study Population | 9 |
| 3.3. | Randomization | 9 |
| 3.4. | Blinding | 9 |
| 3.5. | Study Assessments | 10 |
| 4. | SAMPLE SIZE DETERMINATION | 13 |
| 5. | EFFICACY ENDPOINTS | 13 |
| 5.1. | Primary Endpoints | 13 |
| 5.2. | Secondary Endpoints | 13 |
| 5.3. | Other Safety Endpoint | 13 |
| 5.4. | | 14 |
| 6. | SAFETY ASSESSMENT | 14 |
| 6.1. | Adverse Events | 14 |
| 6.2. | Clinical Safety Laboratory Evaluations | 15 |
| 6.3. | Physical Examinations | 15 |
| 6.4. | Vital Signs, Height, and Weight | 15 |
| 6.5. | | 16 |
| 6.6. | | 16 |
| 7. | ANALYSIS POPULATIONS | 17 |
| 7.1. | Intent-to-Treat Population (ITT) or All Enrolled | 17 |
| 7.2. | Modified ITT Population (mITT) | 17 |
| 7.3. | Per-Protocol (PP) Population | 17 |
| 7.4. | Week 24 Per-Protocol (PP) Population | 17 |
| 7.5. | Safety Population | 17 |

| 8. | STATISTICAL ANALYSIS | 17 |
|--------|----------------------------------------------|----|
| 8.1. | General Statistical Considerations | 17 |
| 8.1.1. | General Analysis Approach | 17 |
| 8.1.2. | | 18 |
| 8.1.3. | Baseline Definition | 19 |
| 8.1.4. | Derived Data | 19 |
| 8.2. | Study Subjects | 19 |
| 8.2.1. | Subject Disposition | 19 |
| 8.2.2. | Protocol Deviations | 20 |
| 8.2.3. | Demographic and Baseline CDI Characteristics | 20 |
| 8.2.4. | Medical and Surgical History | 22 |
| 8.2.5. | Prior and Concomitant Medications | 22 |
| 8.2.6. | Study Drug Compliance | 22 |
| 8.3. | Efficacy Analyses | 22 |
| 8.3.1. | Primary Efficacy Analyses | 22 |
| 8.3.2. | Secondary Efficacy Analyses | 23 |
| 8.3.3. | | 25 |
| 8.3.4. | Subgroup Analyses | 26 |
| 8.4. | Safety Analyses | 27 |
| 8.4.1. | Adverse Events | 27 |
| 8.4.2. | Clinical Laboratory Evaluations | 28 |
| 8.4.3. | Vital Signs | 28 |
| 8.4.4. | Physical Examination | 28 |
| 9. | REFERENCES | 29 |

## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| AE | Adverse event |
|--------------|------------------------------------------------|
| ARB | Antibiotic-resistant bacteria |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body mass index |
| BSS | Bristol Stool Scale |
| C. difficile | Clostridium difficile |
| CDI | Clostridium difficile infection |
| CI | Confidence interval |
| CRE | Carbapenem-resistant Enterobacteriaceae |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DSMC | Data and Safety Monitoring Committee |
| eCRF | Electronic case report form |
| EDC | Electronic Data Capture |
| EIA | Enzyme immunoassay |
| ESBL | Extended-spectrum β-lactamase |
| FMT | Fecal microbiota transplantation |
| GI | Gastrointestinal |
| hCG | Human chorionic gonadotropin |
| ITT | Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-Treat |
| NAP1 | North American Pulse-field type 1 |
| NCI | National Cancer Institute |
| PCR | Polymerase chain reaction |
| PP | Per-Protocol |
| RNA | Ribonucleic acid |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SOC | System Organ Class |
| TEAE | Treatment-emergent adverse event |
| VRE | Vancomycin-resistant enterococci |
| WHO | World Health Organization |

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is created based on Protocol CP101-CDI-E02 (Version 4.0 [Amendment 03], December 20, 2019) and describes in detail the statistical methodology and the statistical analyses to be conducted for the above-mentioned protocol. The SAP will be finalized prior to database lock. Any deviations from this analysis plan will be substantiated by sound statistical rationale and will be documented in the final clinical study report. Changes to the primary efficacy analysis prior to database lock would require an amendment to the protocol and SAP.

#### 2. STUDY OBJECTIVES

The objectives of this Phase 2 open-label study are:

- To evaluate the safety of CP101 treatment in 1) Subjects in PRISM3 who had a CDI recurrence within 8 weeks of receiving CP101 or placebo; OR 2) adults with recurrent CDI who are eligible for direct study entry into PRISM-EXT.
- To evaluate the efficacy of CP101 treatment in 1) Subjects in PRISM3 who had a CDI recurrence within 8 weeks of receiving CP101 or placebo; OR 2) adults with recurrent CDI who are eligible for direct study entry into PRISM-EXT.

#### 3. STUDY DESIGN

#### 3.1. General Study Design and Plan

This open-label extension study entitled PRISM-EXT is evaluating the safety and efficacy in reducing recurrence of CDI in 1) subjects who were enrolled in PRISM3 and had a CDI recurrence within 8 weeks after receipt of CP101 or placebo; OR 2) adults with recurrent CDI who are eligible for direct study entry into the PRISM-EXT study. Subjects who experienced recurrent CDI will undergo screening procedures. Subjects who meet eligibility criteria will be administered CP101.

. The primary efficacy and safety endpoints will be evaluated at 8 weeks post treatment, and all subjects will continue to be followed for an additional 16 weeks for safety and recurrence of CDI.

To qualify for the study, subjects must either have:

1. Previously enrolled in PRISM3, had a CDI recurrence within 8 weeks of receiving CP101 or placebo, and have completed their PRISM3 end of study visit. The definition of recurrent CDI for subjects previously enrolled in PRISM3 is: a) diarrhea (> 3 unformed stools [Bristol Stool Scale score of 6 or 7] per day) for 2 or more consecutive days; b) a stool specimen testing positive for *Clostridium difficile* (*C. difficile*) by the testing algorithm; and c) requiring a course of standard-of-care CDI antibiotics. Additionally, to qualify, recurrent CDI subjects must have received standard-of-care CDI antibiotics for the most recent CDI recurrence (for 10-42 days, with exact duration, antibiotic type, and dose at the discretion of the Investigator) and have an adequate clinical response, defined as ≤ 3

unformed stools in 24 hours for 2 or more consecutive days during standard-of-care CDI antibiotics prior to Treatment.

#### OR

2. Recurrent CDI eligible for direct study entry. Recurrent CDI for direct entry is defined as: a) ≥ 2 episodes of CDI occurring within the previous 6 months (inclusive of the current episode); b) received standard-of-care CDI antibiotics for the most recent CDI episode (for 10-42 days, with exact duration, antibiotic type, and dose at the discretion of the Investigator); c) have an adequate clinical response, defined as ≤3 unformed stools in 24 hours for 2 or more consecutive days during standard-of-care CDI antibiotics prior to treatment.

Subjects who failed screening for the PRISM3 study may be re-evaluated for enrollment into PRISM-EXT if screening criteria are met.

Figure 1. Study Design



CDI = Clostridium difficile infection.

The primary clinical outcomes are safety and prevention of recurrence of CDI. Recurrent CDI is defined as a) diarrhea (> 3 unformed stools [Bristol Stool Scale (BSS) score of 6 or 7] per day) for 2 or more consecutive days; AND b) a stool specimen testing positive for *C. difficile* by a testing algorithm (see Figure below****); AND c) requiring a course of standard-of-care CDI antibiotics. Secondary outcomes include assessment of decolonization of antibiotic-resistant bacteria (ARB)



After the Treatment visit, subjects will return to the clinic at Weeks 8 and 24 for safety and efficacy assessments. Telephone contact, including concomitant medication and adverse event reporting, will occur after the Screening visit, and at Weeks 1, 7, and 23.

Subjects will be issued a paper Memory Aid at the time of informed consent and given training on its use in order to aid in capturing the following information: occurrence of gastrointestinal (GI) symptoms, frequency of stools, fecal urgency, stool incontinence, BSS, and any new medications taken (including antibiotics for treatment of CDI). Subjects will return the Memory Aid to the clinic and will review it with the coordinator at the Screening visit and Treatment (Day 1) after drug administration. At the Week 1 telephone call, the Memory Aid data will be discussed, and subjects will be reminded to bring it to the Week 8 visit. In the event of suspected CDI recurrence, the Memory Aid recorded after Week 1 will be discussed at unscheduled visit(s).

Clinical signs and symptoms of recurrent CDI, including frequency and consistency of stools, will be confirmed by a C. difficile stool testing algorithm. North American Pulse-field type 1 (NAP1)/BI/027 subtyping will be performed if symptoms are consistent with recurrent CDI.



Safety will be assessed via adverse event monitoring, concomitant medication use, physical examinations, vital signs, clinical safety laboratory evaluations, and pregnancy testing (if female is of childbearing potential).

If a subject discontinues from the study early, the subject will be asked to return to the clinic within 14 days after discontinuation to undergo the scheduled Week 24 assessments prior to study discharge. All other subjects will have their final visit at Week  $24 \pm 14$  days.

#### 3.2. Study Population

Approximately 200 subjects 18 years of age or older with either 1) recurrent CDI in PRISM3, and who respond to a standard-of-care CDI antibiotic regimen for the most recent CDI episode, OR 2) recurrent CDI who are eligible for direct study entry, will be administered CP101.

#### 3.3. Randomization

Not applicable. This is an open-label study.

#### 3.4. Blinding

Not applicable. This is an open-label study.

### 3.5. Study Assessments

Table 1 presents the schedule of observations.

Table 1. Schedule of Observations

| | | Screening <sup>1</sup> | Treat.<br>Visit <sup>2</sup> | Efficacy and Safety Assessment Period | | Safety and CDI Recurrence Follow-Up Period | | |
|---|---|---|---|---|---|---|---|---|
| Study time point/activities | Week | Prior to study<br>drug<br>(On-Site) | 0<br>(On-<br>Site) | 1<br>(Tel <sup>9</sup> ) | 7<br>(Tel <sup>9</sup> ) | 8<br>(On-<br>Site) | 23<br>(Tel <sup>9</sup> ) | Week 24 or early<br>termination<br>visit <sup>3</sup><br>(On-Site) |
| | Day | | 1 | 7 ± 2 | 49 ± 3 | 56 ± 3 | 161 ± 7 | 168 ± 14 |
| Screening/Administrative Ass | essments | 5 | | | | | | |
| Informed consent <sup>4</sup> | | X | | | | | | |
| Inclusion/Exclusion Criteria | | X | X <sup>5</sup> | | | | | |
| Demographics | | X | | | | | | |
| Medical history (including BM | )6 | x | | | | | | |
| Memory Aid data recording <sup>7, 8</sup> | | x | Х | X | < | | — (X) <sup>8</sup> —— | > |
| Telephone contact | | X <sup>1</sup> | | X <sub>9</sub> | X <sup>9</sup> | | X <sub>9</sub> | |
| Start/continue treatment of st of-care CDI antibiotics <sup>10</sup> | andard- | х | | | | | | |
| | | x | X <sup>5,11</sup> | | | Х | | X |
| Study drug administration | | | X <sup>12,13</sup> | | | | | |
| Safety Assessments | | | | | | | | |
| Complete physical examination | n <sup>14</sup> | | X <sup>5</sup> | | | | | |
| Symptom-directed physical examination <sup>8,15</sup> | | х | | | | х | | Х |
| Vital signs <sup>8,16</sup> , height <sup>17</sup> , and weight <sup>8,18</sup> | | x | X <sup>19</sup> | | | X | | X |
| Clinical safety laboratory evaluations <sup>20</sup> | | x | X <sup>5</sup> | | | Х | | |
| Drug screen (as needed) <sup>21</sup> | | x | | | | | | |
| Pregnancy testing <sup>22</sup> | | x | X <sup>5</sup> | | | Х | | X |
| Concomitant medications <sup>8,23</sup> | | x | X <sup>5</sup> | < | <> | | | > |
| Adverse events <sup>8,23</sup> | | x | X <sup>23</sup> | <> | | | > | |
| Stool Assessments | | | | | | | | |
| Stool sample collection <sup>8,23</sup> | | Х | X <sup>5,12</sup> | (X) | (X) | х | (X) | х |
| Bristol Stool Scale <sup>8</sup> | | Х | X <sup>5</sup> | Х | (X) | Х | (X) | х |
| | | Х | X <sup>5</sup> | (X) | (X) | Х | (X) | х |
| Assessment for ARB <sup>8,25</sup> | | Х | X <sup>5</sup> | (X) | (X) | х | (X) | Х |
| NAP1/BI/027 subtyping <sup>8</sup> | | | | (X) | (X) | (X) | (X) | (X) |
| C. difficile stool testing algorith | nm <sup>8</sup> | Х | | (X) | (X) | (X) | (X) | (X) |

ARB = antibiotic-resistant bacteria; BMI = body mass index; *C. difficile = Clostridium difficile*; CDI = *Clostridium difficile* infection; GI = gastrointestinal; hCG = human chorionic gonadotropin; NAP1 = North American Pulse-field type 1; Treat. = Treatment; RNA = ribonucleic acid, Tel = telephone assessment.

(X) = in the event of suspected recurrent CDI

1 The Screening visit includes the entire Screening period up to the time of Treatment. The Screening period is limited to 60 days between the signing of informed consent and Treatment. Where referenced as the Screening visit, study-required tests and procedures may be performed on 1 day or across multiple days, but preferably closest to the time of Treatment. During the Screening visit, potential study subjects will be fully informed regarding the nature of the study and possible adverse events and will receive a copy of the informed consent form for review. All subjects must have CDI recurrence defined by the PRISM3 protocol. After the Screening visit, 1 phone call will be made to the subject as a reminder for the upcoming Treatment visit. In the event that the Screening period is planned for > 30 days, additional clinical safety laboratory evaluations may be conducted at the discretion of the Investigator.

| 2 | |
|---|---|
| | . If the subject experiences diarrhea for 2 or more consecutive days during the washout period. |
| | the Investigator should contact the Medical Monitor. |

- 3 If a subject discontinues from the study early, the subject will be asked to return to the clinic within 14 days after discontinuation to undergo the Week 24/End of study assessments prior to study discharge. All other subjects will have their final visit at Week 24 ± 14 days.
- 4 The signing of the informed consent form initiates the screening process. Obtain signed, written informed consent and permission to use Protected Health Information (in accordance with the Health Insurance Portability and Accountability Act). Informed consent must be in place prior to performing any study procedures.
- 5 To be performed prior to study drug administration. NOTE: Missing stool sample does not preclude the subject from Treatment.
- 6 Includes CDI history (e.g., number of prior episodes) and a pre-CDI medically documented weight or BMI (prior to PRISM3) will be obtained.
- 7 Subjects will be issued a paper Memory Aid at the time of informed consent and given training on its use. The Memory Aid data will be discussed at the Screening visit and Treatment visit (Day 1) after drug administration. At Week 1 telephone call, the Memory Aid will be discussed and subjects will be reminded to bring it to the Week 8 visit. Adverse events will be managed according to good clinical practice at the discretion of the treating physician.
- 8 To be performed in the event of a suspected CDI recurrence at the timepoints marked as (X). For stool sample, instructions for at-home stool sample collection, handling, storage, and transportation/shipping are included in the Laboratory Manual and an instruction sheet will be distributed to subjects.
- 9. Subjects will be contacted by telephone. Subjects will be asked about any adverse events, including occurrence of diarrhea. If a subject reports diarrhea, the study staff will review the timing of those episodes and the subject may be asked to submit a stool sample for *C. difficile* testing. Subjects will be asked about their general well-being, changes in their health status, medications, and over-the-counter remedies, and will be reminded about their next study visit. From Screening through study completion, subjects will be reminded to record all signs or symptoms on their Memory Aid, as applicable. If a solicited adverse event is Grade 2 or greater on telephone contact at Week 1, an unscheduled visit will be arranged as soon as possible for evaluation and confirmation of the event. For all subsequent telephone contacts, including Week 7 and Week 23, adverse events will be managed according to good clinical practice at the discretion of the treating physician. Adverse events will be managed according to good clinical practice at the discretion of the treating physician.
  - At Week 8 and 24 visits every effort will be made to conduct an on-site assessment. However, under extenuating subject circumstances that make an on-site visit not feasible and after all reasonable measures to enable the subject's on-site visit have been exhausted, a telephone assessment will be conducted.
- 10 For the most recent CDI episode, the subject will have received standard-of-care CDI antibiotics (10-42 days; with exact duration, antibiotic type, and dose at the discretion of the Investigator).



- 14 A complete physical examination will be performed (including evaluation of general appearance/mental status; head, eyes, ears, nose, throat; and the following body systems: skin, heart, lungs, abdomen, and extremities).
- 15 The Investigator will perform symptom-directed physical examinations based on subjects' signs and symptoms.

- 16 Vital signs (blood pressure, heart rate, and temperature) will be measured per standard of--care. Body temperature should be taken at all visits where vital signs are measured. Vital signs and body temperature should also be measured at time of recurrence, if any.
- 17 Height will be measured at the Screening visit only per standard-of-care.
- 18 Subjects should be weighed per standard-of-care. Height and weight will be used to calculate BMI at Screening, Week 8 and Week 24.
- 19 Vital signs will be measured before and after (within 60 minutes) study drug administration.

  20
- 21 Optional (at the discretion of the Investigator) drug screen includes cotinine (not exclusionary), amphetamines, barbiturates, benzodiazepines, cannabinoids (not exclusionary), cocaine, opioids (not exclusionary), and alcohol.
- 22 Women of childbearing potential enrolled in this study will have serum hCG pregnancy testing administered during Screening and urine pregnancy testing thereafter, at the discretion of the Investigator. Women who are post-menopausal for ≥ 1 year or surgically sterile will not undergo pregnancy testing.
- 23 The adverse event reporting period will begin with informed consent and will continue through study completion or, in the case of withdrawal, until the outcome is determined. Adverse events will be collected after study drug administration on Day 1. Subjects will be asked about any adverse events, including occurrence of diarrhea, at all telephone contact and study visits. If a subject reports diarrhea, the study staff will review the timing of those episodes and the subject may be asked to submit a stool sample for *C. difficile* testing. Subjects will be asked about their general well-being, changes in their health status, medications, and over-the-counter remedies.
- 25 Stool sample collection for the assessment for ARB, defined as vancomycin-resistant enterococci, extended-spectrum β-lactamase organisms, or carbapenem-resistant Enterobacteriaceae, will be performed on samples obtained at Screening, Treatment (Day 1) prior to study drug administration, Week 8, and Week 24. Assessment for ARB may also be performed at any other visit or time point (e.g., time of recurrence, if any).



#### 5. EFFICACY ENDPOINTS

#### **5.1.** Primary Endpoints

The primary endpoints are:

- Incidence of adverse events at through Week 8, and
- Proportion of subjects experiencing sustained clinical cure, defined as absence of recurrent CDI, through Week 8.

#### 5.2. Secondary Endpoints

The secondary endpoints are:

- Proportion of subjects experiencing recurrent CDI through Week 8;
- Proportion of subjects experiencing recurrent CDI with ribosomal NAP1/BI/027 *C. difficile* subtype through Week 8;
- Time-to-first recurrent CDI episode during the study (Day 1 through Week 8);
- Proportion of subjects experiencing sustained clinical cure at Week 24;
- Proportion of subjects experiencing recurrent CDI through Week 24;
- Time-to-first recurrent CDI episode during the study (Day 1 through Week 24);
- Incidence of hospitalization due to recurrent CDI through Week 8 and through Week 24;
- Incidence of decolonization of antibiotic-resistant bacteria (ARB), defined as vancomycin-resistant enterococci, extended-spectrum β-lactamase (ESBL) organisms, or carbapenem-resistant Enterobacteriaceae (CRE) at Week 8 and Week 24 among co-colonized subjects at baseline;
- Change in body mass index (BMI) by Week 8 and Week 24 relative to medically documented pre-CDI BMI; and
- Incidence of newly diagnosed autoimmune disease through Week 8 and Week 24.

#### 5.3. Other Safety Endpoint

The other safety endpoint is:

• Incidence of adverse events through Week 24.



#### 6. SAFETY ASSESSMENT

#### 6.1. Adverse Events

The adverse event reporting period will begin with informed consent and will continue through study completion or, in the case of withdrawal, until the outcome is determined. Adverse events will be assessed at each visit and through telephone contact with the subject. Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, Version 20.1).

The intensity of an adverse event will be graded according to the scale below in addition to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) for Grading the Severity of Adult Adverse Events. The clinical significance of the adverse event is determined by the Investigator.

| Grade | Description |
|---|---|
| Grade 1 (Mild): | Asymptomatic or mild symptoms; clinical or diagnostic |
| Grade 2 (Moderate): | observations only; intervention not indicated<br>Minimal, local or noninvasive intervention indicated;<br>limiting age-appropriate instrumental activities of daily |
| Grade 3 (Severe): | living Medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; |
| Grade 4 (Life-Threatening): | disabling; limiting self-care activities of daily living<br>Life-threatening consequences; urgent intervention<br>indicated |
| Grade 5 (Death): | Death related to adverse event |

In this study, if a subject has CDI recurrence in the study, then CDI will not be recorded as an adverse event; instead, it will be considered an on-study recurrent CDI episode and will be included in the determination of efficacy. If the on-study recurrent CDI episode results in hospitalization of the subject for more than 24 hours, this will be recorded as an SAE and reported per the criteria for safety reporting.

#### 6.2. Clinical Safety Laboratory Evaluations

Samples of blood and urine are scheduled for collection at Screening, at Treatment (Day 1) prior to study drug administration, and at Week 8; specific tests performed at each visit are shown in Table 2. The total volume of blood collected at scheduled study visits will be approximately 123 mL. Additional follow-up samples for clinical laboratory testing should be obtained as clinically indicated. A 3-mL serum aliquot will be collected at each time point and archived for safety testing as may be required by emergence of adverse conditions.

Subjects with a white blood cell count  $\geq 15 \times 10^9$ , laboratory evidence of acute kidney injury, or an absolute neutrophil count of  $< 1 \times 10^9$  neutrophils at Screening are to be excluded from the study.

All clinical laboratory testing, with the exception of optional drug testing or on-site urine pregnancy testing during the treatment period for females of childbearing potential, will be performed by the central clinical laboratory.

Category Analyte Hematology Complete blood count with differential Chemistry Activated partial thromboplastin time, prothrombin time, and international normalized Coagulation Urinalysis Screening only Drug Screen Optional drug screen including cotinine (not exclusionary), amphetamines, barbiturates, benzodiazepines, cannabinoids (not exclusionary), cocaine, opiates (not exclusionary), and (Optional, at discretion of the Investigator) alcohol. Pregnancy Serum hCG for women of childbearing potential.

Table 2. Clinical Laboratory Safety Tests

hCG = human chorionic gonadotropin.

#### 6.3. Physical Examinations

A complete physical examination (including evaluation of general appearance/mental status; head, eyes, ears, nose, throat; and the following body systems: skin, heart, lungs, abdomen, and extremities) will be performed at the time points listed in the Schedule of Observations (Table 1).

The Investigator will perform the symptom-directed physical examinations based on subjects' signs and symptoms at the time points listed in the Schedule of Observations (Table 1).

#### 6.4. Vital Signs, Height, and Weight

Vital signs (blood pressure, heart rate, and temperature) will be assessed per standard-of-care as listed in the Schedule of Observations (Table 1). Vital signs will be measured before and after (within 60 minutes) study drug administration. Body temperature should be taken at all

visits where vital signs are measured. Vital signs and body temperature should also be measured at time of recurrence, if any.

Body weight and height (Screening only) will be measured per standard-of-care (the height will not be re-measured if it has been collected in the PRISM3 trial). Height and weight will be used to calculate BMI. A pre-CDI medically documented weight or BMI will be obtained. BMI will be calculated from weight collected at Week 8 and Week 24 as well.

| 6.5. | |
|------|---|
| | I |
| | _ |
| _ | |
| _ | |
| 6.6. | |

#### 7. ANALYSIS POPULATIONS

All analyses will be performed separately for subjects previously enrolled in PRISM3 and direct entry subjects as well as for both groups combined. For subjects previously enrolled in PRISM3, it will also be summarized by prior exposure (CP101 or placebo) in PRISM3.

Each analysis population includes both rollover subjects from PRISM3 study and subjects with direct entry into the PRISM-EXT study.

#### 7.1. Intent-to-Treat Population (ITT) or All Enrolled

All subjects enrolled into the study.

#### 7.2. Modified ITT Population (mITT)

All subjects in the ITT population who receive at least 1 capsule of study drug at Treatment (Day 1). The mITT population will be the primary analysis population for all efficacy analyses.

#### 7.3. Per-Protocol (PP) Population

All subjects in the mITT population who have received at least 80% of study medication, completed 8 weeks of follow up or had documented CDI recurrence prior to the 8-week follow-up and did not have any major protocol deviation that affect the efficacy of the study drug through the Week 8 Visit.

#### 7.4. Week 24 Per-Protocol (PP) Population

All subjects in the mITT population who have received at least 80% of study medication, completed 24 weeks of follow up or had documented CDI recurrence prior to the 24-week follow-up and did not have any major protocol deviation that affect the efficacy or safety of the study drug. The Week 24 PP Population will be used for all analyses of the Week 24 endpoints where the PP Population is specified.

Based on the above criteria, the validity listings will be provided to identify which subjects to be excluded from the PP Populations. After the study team's review, the decision to exclude a subject from the PP Populations will be finalized and a list of subjects with major protocol deviations leading to exclusion from the PP Populations will be finalized and documented.

#### 7.5. Safety Population

All enrolled subjects who received at least 1 capsule of study drug. Unless otherwise stated, the Safety population will be the default analysis population for all safety analyses.

#### 8. STATISTICAL ANALYSIS

#### 8.1. General Statistical Considerations

#### 8.1.1. General Analysis Approach

• All table summaries and listings will present the results separately for subjects previously enrolled in PRISM3 and direct entry subjects as well as for both groups combined. For

subjects previously enrolled in PRISM3, it will also be displayed by prior exposure (CP101 or placebo) in PRISM3.

- For purposes of all analysis and reporting, days will be numbered relative to the first day of dosing. Day 1 will be defined as the date on which a subject receives the first dose of study drug, as recorded on the electronic case report form (eCRF). The day prior to the first dose of study drug is Day -1;
- Descriptive statistical methods will be used to summarize study data. Unless stated otherwise, the term "descriptive statistics" refers to number of subjects (n), mean, median, standard deviation, minimum, and maximum for continuous data, and refers to frequencies and percentages for categorical data. For categorical data summary, number of subjects with missing data will be included and percentages will be calculated based on the total number of subjects in the specified analysis population. For some data that may be presented as continuous variables, there may be scientific reasons to present those data in constructed categories as well (e.g., BMI). Reasons for the categories will be described in the Clinical Study Report.
- Individual data listings of all data represented on the eCRF will be presented. Sort order for data listings will be subject identification number, visit, and time point where appropriate.
- The SAP will be finalized and approved by signatures and dates prior to database lock. The SAP will take precedence over the protocol for details about the statistical analyses for the study except the primary efficacy analyses which would require a protocol amendment. In addition to the analyses specified in the SAP, other exploratory analyses and graphical representations of the results may be produced after review of the data (post-hoc).
- Verbatim terms recorded for medical history conditions, surgical history procedures, and adverse events will be mapped to a SOC and preferred term using MedDRA, and all prior and concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary (B3 September 2018).

| 8.1.2. |
|--------|



#### **8.1.3.** Baseline Definition

For all efficacy and safety endpoints, baseline is defined as the last measurement or assessment prior to the administration of study drug in the extension study.

#### 8.1.4. Derived Data

- Age will be calculated using the subject's date of birth and the date the subject signed informed consent [integer part of (informed consent date birth date)/365.25].
- Change from baseline values will be calculated as the value at a post-baseline time point minus the baseline value.
- The Day on which an AE occurrence is noted will be calculated relative to the date of the first dose of study drug; Day = (date of AE date of first dose) if date of AE is before date of first dose, Day = (date of AE date of first dose + 1) if date of AE is on or after date of first dose.
- Other derived variables summarized in tables (with individual values provided in listings) will be described in footnotes of the tables where appropriate.

The detailed derivation for the efficacy and safety data will be documented in a separate derived datasets specification.

#### 8.2. Study Subjects

#### 8.2.1. Subject Disposition

The number of subjects who are enrolled, treated, complete the study, and discontinue from the study will be summarized for the ITT population. Subject disposition will also be summarized by study site.





In addition, the total number of subjects for each defined population will be tabulated. Reasons for exclusions from analyses populations will be tabulated.

#### **8.2.2.** Protocol Deviations

The number of subjects with at least one reportable protocol deviation, and the number of subjects with at least one reportable deviation in each deviation category defined in the study protocol deviation plan will be presented based on the ITT and mITT populations. In addition, the protocol deviations related to COVID-19 pandemic will be categorized and summarized separately.

Protocol deviations will also be listed by subject.

#### 8.2.3. Demographic and Baseline CDI Characteristics

The following demographics will be summarized:

- Age (years) and age categorized as <65 vs.  $\ge65$  years, and <70, 70-79, or  $\ge80$  years;
- Sex;
- Race;
- Ethnicity;
- Pre-CDI weight (kg);
- Height (cm);
- Pre-CDI BMI (kg/m<sup>2</sup>);

• Charlson comorbidity index  $(CCI)^1$  and CCI categories (<3 and  $\geq$ 3).

The following baseline CDI characteristics will be summarized:

- CARDS score<sup>2</sup> and score categories (<5, 5-9, 10-14, and  $\ge$ 15);
- GEIH-CDI score<sup>3</sup> and score categories ( $\leq 3$  and  $\geq 3$ );
- Previous CDI-associated hospitalizations (0, 1, 2, 3+, and 1+);
- Previous CDI episodes
  - Total number of CDI episodes in previous 6 months (inclusive of the current episode) (1, 2, 3, and >3)



Demographic and baseline characteristics will be summarized with descriptive statistics or counts and percentages of subjects as appropriate in all analysis populations.

#### 8.2.4. Medical and Surgical History

Medical and surgical history terms will be coded using MedDRA (Version 20.1). Medical and surgical history will be summarized and MedDRA SOC and preferred term in all analysis populations.

All Medical and surgical history will be listed by subject.

#### 8.2.5. Prior and Concomitant Medications

Prior and concomitant medications will be coded using the WHO Drug Dictionary (B3 September 2018). Prior medications will include medications used before the administration of study drug. Any medications used on or after the administration of study drug will be included as concomitant medications.

The number and percentage of subjects taking prior medications will be summarized in all analysis populations by Anatomical Therapeutic Chemical (ATC) class and preferred term.

The number and percentage of subjects taking concomitant medications will be summarized in the same manner.

All prior and concomitant medications and procedures will be listed by subject.

#### 8.2.6. Study Drug Compliance

In addition, summary tables will be provided to show the number and percentage of subjects with compliance in the following categories: <80% and  $\ge80\%$ .

#### 8.3. Efficacy Analyses

#### 8.3.1. Primary Efficacy Analyses

The primary efficacy endpoint is defined as the proportion of subjects with sustained clinical cure (Table 3) through Week 8 calculated as the number of subjects with sustained clinical cure through Week 8 divided by the total number of subjects in the analysis population.





The proportion of subjects with sustained clinical cure through Week 8 will be summarized in the mITT population, separately for subjects previously enrolled in PRISM3 and direct entry subjects as well as for both groups combined. For subjects previously enrolled in PRISM3, it will also be summarized by prior exposure (CP101 or placebo) in PRISM3. The proportion will be presented together with 95% exact binomial confidence intervals (CIs).

#### 8.3.2. Secondary Efficacy Analyses

#### Proportion of subjects with sustained clinical cure through Week 8 in the PP Population

Proportion of subjects with sustained clinical cure through Week 8 will be summarized for the PP Population. The proportion will be presented together with 95% exact binomial CIs.

# <u>Proportion of subjects experiencing recurrent CDI through Week 8 by ribosomal NAP1/BI/027 subtype at CDI recurrence</u>

The proportion of subjects experiencing recurrent CDI at Week 8 will be summarized by ribosomal NAP1/BI/027 *C. difficile* subtype at CDI recurrence for the mITT and PP populations within each subtype (NAP1/BI/027 vs. not NAP1/BI/027). The proportion will be presented together with 95% exact binomial CIs.



#### **Proportion of subjects experiencing CDI Recurrence at Week 8**

The proportion of subjects with CDI recurrence through Week 8 will be summarized in the mITT and PP population, separately for subjects previously enrolled in PRISM3 and direct entry subjects as well as for both groups combined. For subjects previously enrolled in PRISM3, it will also be summarized by prior exposure (CP101 or placebo) in PRISM3. The proportion will be presented together with 95% exact binomial confidence intervals (CIs).

#### Proportion of subjects experiencing sustained clinical cure at Week 24

The proportion of subjects experiencing sustained clinical cure through Week 24 is defined as the number of subjects with sustained clinical cure through Week 24 divided by the total number of subjects in the analysis population. Investigator reported suspected CDI recurrence will be adjudicated by an independent Adjudication Board in a blinded fashion prior to database lock. The determination of "sustained clinical cure" is defined in Table 4. The proportion of subjects experiencing sustained clinical cure at Week 24 will be summarized by for the mITT and PP populations. The proportions will be presented together with 95% exact binomial confidence intervals.



#### Proportion of subjects experiencing CDI Recurrence at Week 24

The proportion of subjects experiencing CDI recurrence through Week 24 is defined as the number of subjects with CDI recurrence through Week 24 divided by the total number of subjects in the analysis population. Investigator reported suspected CDI recurrence will be adjudicated by an independent Adjudication Board in a blinded fashion prior to database lock for Week 24 and will constitute the determination of "CDI recurrence" as defined in column 4 of Table 4. The proportion of subjects experiencing CDI Recurrence at Week 24 will be

summarized for the mITT and PP populations. The proportion will be presented together with 95% exact binomial CIs.

#### Incidence of hospitalization due to recurrent CDI through Week 8 and Week 24

Incidence of hospitalization (including emergency room visits) due to recurrent CDI is defined as the number of subjects who were hospitalized due to recurrent CDI divided by the total number of subjects in the analysis population. Incidence of hospitalization due to recurrent CDI at Week 8 and Week 24 will be summarized for the mITT and PP populations. The proportion will be presented together with 95% exact binomial CIs. In addition, duration of hospitalization will be summarized for the mITT and PP populations. Duration of hospitalization is calculated as the total number of days of hospitalization.

#### **Incidence of decolonization of ARB at Week 8 and Week 24**

Incidence of decolonization of ARB is defined as the number of subjects who experienced decolonization of ARB (VRE, ESBL organisms, or CRE) divided by the total number of subjects with ARB at baseline in the analysis populations. Incidence of decolonization of ARB at Week 8 and Week 24 will be summarized for the mITT and PP populations. The proportion will be presented together with 95% exact binomial CIs.

| Change in BMI at Week 8 and Week 24 |
|---|
| Change from pre-CDI BMI will be calculated at the specified study visit as the value at the specified study visit minus the pre-CDI value. Change in BMI at Week 8 and Week 24 relative to medically documented pre-CDI BMI will be summarized in the mITT and PP populations. |
| 8.3.3. |



#### 8.3.4. Subgroup Analyses

The following subgroups based on baseline characteristics will be used for subgroup analyses for the primary efficacy endpoint in the mITT and PP populations.

- Age group (<65 years vs. ≥65 years)
- Age group ( $<70, 70-79, \text{ and } \ge 80 \text{ years}$ )
- Gender group (male vs. female)
- Race group (Caucasian vs. others)
- Charlson Comorbidity Index (<3 vs. ≥3)
- CARDS score ( $<5, 5-9, 10-14, and \ge 15$ )
- GEIH-CDI score ( $\leq 3 \text{ vs.} > 3$ )
- Previous CDI episodes total number of CDI episodes in previous 6 months (1, 2, 3, and >3)
- Previous CDI-associated hospitalizations (Yes vs. No)





Ad-hoc Analyses

Additional analyses may be performed and will be considered as ad-hoc analyses and exploratory in nature.

#### 8.4. Safety Analyses

All safety summaries and analyses will be performed on the Safety population. All subjects will be summarized according to the treatment actually received.

Safety will be evaluated by presenting summaries of AEs, vital signs, laboratory evaluations and physical examinations. For each safety parameter, unless otherwise stated, the last assessment made prior to the administration of study drug will be used as the baseline value for all analyses.

#### **8.4.1.** Adverse Events

Any event reported on the eCRF that occurs during or after the administration of study drug is defined as treatment-emergent adverse event (TEAE). Additionally, it will be assumed that an adverse event that was reported to have started at Treatment (Day 1) without an associated onset time may have occurred after the administration of study drug. Hence, adverse events occurring at Treatment (Day 1) with no associated onset time are assumed to be treatment-emergent.

For the primary safety endpoint, the incidence rate of TEAEs will be presented through Week 8.

For the other safety endpoints, the incidence rate of TEAE will be presented through Week 24.

In addition, an overview of TEAEs will be provided which summarizes the incidence of the following information:

- All TEAEs
- Drug-related TEAEs
- Maximum severity of TEAEs
- Deaths

#### • Serious adverse events (SAEs)

The number and percentage of subjects who experienced at least one TEAE will be presented by system organ class and preferred term. Drug-related TEAEs, withdrawals due to TEAEs, and all SAEs will be summarized in the same manner.

Although a subject may have two or more TEAEs, the subject is counted only once within a System Organ Class and Preferred Term category. The same subject may contribute to two or more preferred terms in the same System Organ Class category.

A list of subjects who have SAEs, and a list of subjects who discontinue from study drug will be provided. All adverse events will be listed.

Newly diagnosed autoimmune disease will be reported as an AE. Newly diagnosed autoimmune disease is defined autoimmune disease occurs on or after the administration of study drug. Incidence of newly diagnosed autoimmune disease at Week 8 and Week 24 will be summarized for the Safety population. The number and percentage of subjects who experienced treatment-emergent autoimmune disease will be presented by system organ class and preferred term.

The solicited signs and symptoms collected will be entered in the eCRF and will be graded for severity. The number and percentage of subjects who experienced solicited signs and symptoms will be presented by severity at baseline and post-baseline maximum severity.

#### **8.4.2.** Clinical Laboratory Evaluations

Descriptive statistics for clinical laboratory tests for hematology, chemistry, and coagulation listed in Table 2 will be presented by study visit as well as the change from baseline.

Laboratory abnormalities will be graded according to NCI CTCAE Version 4.03 (for analytes where CTCAE grading applies). The number and percentage of subjects experiencing treatment-emergent graded toxicities will be summarized by severity grade. A shift table, presenting the 2-way frequency tabulation for baseline and the worst post-treatment value according to the NCI-CTCAE grade, will be provided. For laboratory parameters with no CTCAE grading, shift tables (with categories of low, normal, high) from baseline to worst post-treatment value will be provided. Both scheduled and unscheduled post-treatment values during the treatment period will be considered.

All clinical laboratory data will be listed. Values outside the normal ranges will be identified in the data listings with flags for low (L) and high (H).

#### 8.4.3. Vital Signs

Descriptive statistics for vital signs (temperature, heart rate, blood pressure and respiratory rate) will be presented by study visit and for the change from baseline. Descriptive statistics for weight will be presented by study visit and for the change from pre-CDI weight.

A listing of all vital signs will be provided by subject.

#### **8.4.4.** Physical Examination

Physical examination findings will be summarized for any abnormal findings that are considered clinically significant in the opinion of the Investigator. These will be recorded as

adverse events or be captured on the medical history if they are already present during Screening.

Physical examination findings will be listed by subject.

#### 9. REFERENCES

- 1. Charlson comorbidity index with age-adjustment (Suidan et al. Gynecol Oncol. 2015; 138(2):236-251;
- 2. C. difficile Associated Risk of Death Score (CARDS) (Kassam et al. Aliment Pharmacol Ther. 2016; 43(6):725-733;
- 3. GEIH-CDI score (Cobo et al. Int J Antimicrob Agents. 2018; 51(3):393-398.